CLINICAL TRIAL: NCT03330743
Title: Parent Mentor Interventions for Early Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Byron A Foster, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00017356
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention)
- Parent Mentor (Placebo Comparator)
  Interventions: Behavioral: Parent Mentor with Standard Education
- Parent Mentor with Positive Deviance (Active Comparator)
  Interventions: Behavioral: Parent Mentor with Positive Deviance

INTERVENTIONS:
Behavioral: Parent Mentor with Standard Education — Parent mentors will provide coaching based on the current guidelines around diet and physical activity
  Arms: Parent Mentor
Behavioral: Parent Mentor with Positive Deviance — Parent mentors will provide coaching based on findings from the positive deviance study
  Arms: Parent Mentor with Positive Deviance

SUMMARY:
The purpose of this clinical trial is to identify the most effective strategy for intervention to change behaviors and affect weight status in obese children 2-5 years of age within the context of early childhood education centers.

DETAILED DESCRIPTION:
The primary aim is to test an intervention to disseminate and promote the adoption of positive deviance behaviors among parents of obese Hispanic children using peer mentors. This trial will evaluate the efficacy and feasibility of this approach in reducing adiposity among a high-risk population of children.

Our central hypothesis is that children randomized to the intervention with a parent mentor using positive deviance methods with have a greater reduction in adiposity as measured by body mass index (BMI) compared with a parent mentor using traditional education or a control receiving usual education.

ELIGIBILITY:
Inclusion Criteria:

* 2-5 years of age child, Hispanic ethnicity, attends the Head Start facility

Exclusion Criteria:

* any major medical disorder impairing growth or development

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
BMIz | 6 months post-enrollment
  standardized BMI for age and sex

SECONDARY OUTCOMES:
Self-efficacy | 6 months post-enrollment
  Parenting self-efficacy around specific topics

CONTACTS AND LOCATIONS:
Overall Officials: Byron Foster, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Foster BA, Alvarez HO, Padilla T, Meyer JS. Longitudinal Examination of Hair Cortisol Concentrations and Weight Changes in Preschool-Aged Children of Latino Farmworkers. Child Obes. 2023 Sep;19(6):399-407. doi: 10.1089/chi.2022.0103. Epub 2022 Aug 24. PMID 36036733
- [Derived] Foster BA, Weinstein K, Padilla T, Martinez C, Angeles-Ramos D. Growing Healthy Together: A Randomized Clinical Trial Using Parent Mentors for Early Childhood Obesity in Low-Income, Latino Families. Child Obes. 2022 Apr;18(3):168-177. doi: 10.1089/chi.2021.0165. Epub 2021 Oct 5. PMID 34613828
- [Derived] Foster BA, Weinstein K, Shannon J. Growing Healthy Together: protocol for a randomized clinical trial using parent mentors for early childhood obesity intervention in a Latino community. Trials. 2019 Apr 25;20(1):235. doi: 10.1186/s13063-019-3342-3. PMID 31023345